CLINICAL TRIAL: NCT03923309
Title: Oncologic Risk of Rectal Preservation Against Medical Advice After Chemoradiotherapy for Rectal Cancer: a Multicenter Comparative Study With Rectal Preservation as Supported by Surgeon
Brief Title: Oncologic Risk of Rectal Preservation Against Medical Advice After Chemoradiotherapy for Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Cancer Center, Korea (Other Government); Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Sung-Bum Kang, Colorectal Surgeon, University Professor, Seoul National University Hospital
Other Study IDs: B-1711/433-102
Record Dates: First submitted 2019-04-16; First posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Rectal Cancer; Chemoradiation
Keywords: Organ preservation; Oncologic outcome
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intended rectal preservation: When rectal preservation (non-operative management or local excision) was agreed by their surgeon.
- Unintended rectal preservation: When rectal preservation (non-operative management or local excision) was disagreed by their surgeon.

SUMMARY:
Though refusal of radical surgery was often happened in rectal cancer patient after neoadjuvant chemoradiotherapy, little is currently known about the actual oncologic outcome of it. Thus the investigators designed this study to compare the oncologic outcome of unintended rectal preservation with intended rectal preservation by surgeon.

DETAILED DESCRIPTION:
The investigators identified patients whose organ were preserved by non-operative management or local excision after neoadjuvant chemoradiotherapy for mid to low rectal cancer. Then, the patients were categorized into two groups according to the agreement on omitting radical surgery (rectal preservation). When treatment decision was agreed by their surgeon, the patients were categorized as intended rectal preservation. When there was disagreement by surgeon on rectal preservation, then the patients categorized as unintended rectal preservation. Oncologic outcome was compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

* biopsy proven rectal cancer (anal verge ≤ 10cm)
* neoadjuvant radiotherapy or chemoradiotherapy
* no radical surgery after neoadjuvant therapy

Exclusion Criteria:

* other malignant disease
* other fatel disease
* incompletion of half of radiotherapy course
* metastasis on initial presentation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Intended organ preservation
  * non-operative management or local excision selected by surgeon
  Unintended organ preservation
  * non-operative management or local excision persisted by patient and disagreed by surgeon
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
3-year overall survival | from date of completion of chemoradiotherapy until the date of death from any cause, whichever came first, assessed at 31th December 2017 by checking expire date of a resident registration number
  Overall survival rate at 3-year after completion of chemoradiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Hwan Oh, Ph.D., Principal Investigator — National Cancer Center, Korea; Kyu Joo Park, Ph.D., Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - National Cancer Center, Korea, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No
The row data generated during and/or analysed during the current study couldn't be shared to public or other researcher because of institutional policy.

REFERENCES:
- [Background] Ellis CT, Samuel CA, Stitzenberg KB. National Trends in Nonoperative Management of Rectal Adenocarcinoma. J Clin Oncol. 2016 May 10;34(14):1644-51. doi: 10.1200/JCO.2015.64.2066. Epub 2016 Mar 28. PMID 27022115
- [Background] Cassidy RJ, Switchenko JM, Cheng E, Jiang R, Jhaveri J, Patel KR, Tanenbaum DG, Russell MC, Steuer CE, Gillespie TW, McDonald MW, Landry JC. Health care disparities among octogenarians and nonagenarians with stage II and III rectal cancer. Cancer. 2017 Nov 15;123(22):4325-4336. doi: 10.1002/cncr.30896. Epub 2017 Jul 31. PMID 28759121
- [Background] Lee DY, Teng A, Pedersen RC, Tavangari FR, Attaluri V, McLemore EC, Stern SL, Bilchik AJ, Goldfarb MR. Racial and Socioeconomic Treatment Disparities in Adolescents and Young Adults with Stage II-III Rectal Cancer. Ann Surg Oncol. 2017 Feb;24(2):311-318. doi: 10.1245/s10434-016-5626-0. Epub 2016 Oct 20. PMID 27766558